CLINICAL TRIAL: NCT01071798
Title: A Prospective, Multi-center, Non-interventional Observational Study to Evaluate the Safety and Effectiveness of MabThera® (Rituximab) Within the First 6 Months (in Case of Re-therapy the First 12 Months) of Treatment in Patients With Severe Active Rheumatoid Arthritis in Routine Care
Brief Title: An Observational Study on the Safety and Effectiveness of Rituximab in Patients With Severe Active Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22639
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Main Analysis Set: Participants who received at least one cycle of rituximab
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — As prescribed by physician
  Other Names: Mabthera; Rituxan

SUMMARY:
This prospective observational study aims to evaluate safety, application and onset of effect of rituximab in clinical routine treatment of severe active rheumatoid arthritis during the first 6 months (in case of re-therapy: 12 months).

ELIGIBILITY:
Inclusion Criteria:

* No pretreatment with rituximab
* Age 18 years or older
* Patients with active, severe rheumatoid arthritis with prescription of rituximab according to German Summary of Product Characteristics (SmPC - "Fachinformation")
* Patients with signed informed consent
* Female patients with secure contraception

Exclusion Criteria:

* Violation of Selection criteria:

  1. Active severe infection
  2. Severe heart failure (NYHA class IV) or severe, uncontrollable heart disease
  3. Participation in an interventional study within the last 3 months before therapy start with rituximab
  4. Pretreatment with rituximab
  5. Age <18 years
  6. Known intolerability of monoclonal antibodies or chimeric monoclonal antibodies
  7. Known pregnancy or breastfeeding
* Data of patients without approval of data by the physician
* Patients without informed consent
* Double documentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants starting treatment with rituximab
Sampling Method: Probability Sample
Enrollment: 1653 (Actual)
Dates: Start 2010-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Berlin, Germany

REFERENCES:
- [Result] Tony HP, Roll P, Mei HE, Blumner E, Straka A, Gnuegge L, Dorner T; FIRST/ ReFIRST study teams. Combination of B cell biomarkers as independent predictors of response in patients with rheumatoid arthritis treated with rituximab. Clin Exp Rheumatol. 2015 Nov-Dec;33(6):887-94. Epub 2015 Oct 30. PMID 26517829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data were recorded throughout Germany in 264 study centers.
Period: Participants Who Received One Cycle
Arm/Group | Main Analysis Set
Started | 1653
Baseline and Safety Analysis Set | 1653
Completed | 1588
Not Completed | 65
Not completed — Lack of Efficacy | 18
Not completed — Lack of tolerability | 14
Not completed — Patient requirement | 20
Not completed — Death | 5
Not completed — Change of therapy | 6
Not completed — Severe concomitant disease | 2
Period: Subpopulation Who Received Two Cycles
Arm/Group | Main Analysis Set
Started | 820
Baseline and Safety Analysis Set | 820
Completed | 805
Not Completed | 15
Not completed — Remission | 1
Not completed — Lack of Efficacy | 3
Not completed — Lack of Tolerability | 4
Not completed — Patient Requirement | 7

BASELINE CHARACTERISTICS:
Population: Main analysis population
Arm/Group | Main Analysis Set
Number analyzed (Participants) | 1653
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.0 [52.0 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1199
  Male | 454

OUTCOME MEASURES:

1. Primary Outcome: DAS28 Score
Description: The DAS28 consists of swollen joint count (SJC) and tender joint count (TJC) measurements, the erythrocyte sedimentation rate (ESR) in millimeters per hour (mm/hr), and the Patient's Global Assessment of Disease Activity (participant-rated rheumatoid arthritis [RA] activity assessment) with transformed scores ranging 0 to 10; higher scores indicate greater affectation due to disease activity.
Time Frame: at baseline of each cycle and approximately 15 days, 6 weeks (only cycle 1), 12 weeks (3 months), 18 weeks (only cycle 1), and 24 weeks (6 months) after the start of the respective cycle
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Seronegative Participants: Subgroup of seronegative participants
- Seropositive Participants: Subgroup of seropositive participants
Arm/Group | Main Analysis Set | Seronegative Participants | Seropositive Participants
Number analyzed (Participants) | 1653 | 150 | 1186
units on a scale
  Baseline (n=1396,150,1186) | 5.3 (1.4) | 5.0 (1.4) | 5.4 (1.4)
  15 days (n=1133,120,957) | 4.8 (1.4) | 4.6 (1.4) | 4.9 (1.4)
  6 weeks (n=778,73,670) | 4.4 (1.4) | 4.3 (1.4) | 4.4 (1.4)
  12 weeks (n=785,75,666) | 4.0 (1.3) | 4.0 (1.3) | 4.0 (1.3)
  18 weeks (n=601,57,520) | 3.8 (1.3) | 4.1 (1.4) | 3.8 (1.3)
  24 weeks (n=641,60,553) | 3.8 (1.4) | 4.1 (1.3) | 3.8 (1.4)
  Start 2nd cycle (n=588,47,517) | 4.1 (1.4) | 4.2 (1.5) | 4.1 (1.4)
  15 days (n=525,43,460) | 3.9 (1.4) | 4.0 (1.5) | 3.8 (1.4)
  3 months (n=451,37,393) | 3.5 (1.3) | 3.7 (1.5) | 3.5 (1.3)
  6 months (n=491,34,438) | 3.5 (1.4) | 3.9 (1.6) | 3.5 (1.3)

2. Primary Outcome: HAQ Disability Index (HAQ-DI)
Description: The HAQ-DI score consists of questions referring to 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. For each of the categories, participants reported the amount of difficulty they had in performing 2 or 3 specific subcategory items. The standard disability score is calculated from the 8 categories by dividing the sum of the individual categories by the number of categories answered, yielding a score from 0 (without any difficulty) to 3 (unable to do).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Analysis Set | Seronegative Participants | Seropositive Participants
Number analyzed (Participants) | 1653 | 174 | 1326
units on a scale
  Baseline (n=1579,174,1326) | 1.5 (0.7) | 1.5 (0.7) | 1.5 (0.7)
  15 days (n=1514,169,1270) | 1.4 (0.7) | 1.4 (0.8) | 1.4 (0.7)
  6 weeks (n=983,0,0) | 1.3 (0.7) | NA (NA) — These data were not collected | NA (NA) — These data were not collected
  12 weeks (n=1015,116,848) | 1.2 (0.7) | 1.3 (0.8) | 1.2 (0.7)
  18 weeks (n=784,0,0) | 1.2 (0.7) | NA (NA) — These data were not collected | NA (NA) — These data were not collected
  24 weeks (n=810,90,681) | 1.2 (0.7) | 1.3 (0.8) | 1.2 (0.7)
  Start 2nd cycle (n=768,68,669) | 1.2 (0.7) | 1.4 (0.8) | 1.2 (0.7)
  15 days (n=706,67,610) | 1.2 (0.7) | 1.2 (0.7) | 1.2 (0.7)
  3 months (n=594,59,508) | 1.1 (0.7) | 1.3 (0.7) | 1.1 (0.7)
  6 months (n=626,56,546) | 1.2 (0.7) | 1.3 (0.8) | 1.1 (0.7)

3. Secondary Outcome: Percentage of Participants With a Treatment-Emergent Adverse Event (TEAE)
Time Frame: during Cycle 1, during Cycle 2, during the trial (within 12 months)
Measure: Number; unit: percentage of participants
Groups:
- Cycle 1: During Cycle 1 - Main Analysis Set
- Cycle 2: During Cycle 2 - Subpopulation With Two Cycles
- Total: During the Trial - All Participants
Arm/Group | Cycle 1 | Cycle 2 | Total
Number analyzed (Participants) | 1653 | 820 | 1653
percentage of participants
  Any TEAE | 28.5 | 21.1 | 34.8
  Any serious TEAE | 8.7 | 5.7 | 10.9
  Any related TEAE | 6.1 | 6.2 | 8.5
  Any related serious TEAE | 2.5 | 1.3 | 3.0
  Any severe TEAE | 5.5 | 4.3 | 7.0
  Any TEAE leading to discontinuation | 1.9 | 1.3 | 2.6
  Any TEAE leading to death | 0.5 | 0.2 | 0.6

4. Secondary Outcome: Number of Participants Who Received Only One Treatment Cycle With Clinically Relevant Changes in HAQ-Score at Last Visit During Therapy Compared to Baseline (Categorized)
Description: In the Main Analysis Set participants with only one treatment cycle, the HAQ score was categorized for 12 subgroups as Clinically relevant improvement of HAQ-Score ≥0.3, Other or no clinical relevant change of HAQ Score, or Clinically relevant worsening of HAQ Score ≥0.3. Subgroups are defined as Anti-Cyclic citrullinated peptide (CCP) and Rheumatoid factor (RF) negative (-), positive (+), or Non-specified (n.sp.) and Seropositive Non-specified (n.sp.), Seronegative, or Seropositive.
Time Frame: 24 weeks after starting Cycle 1
Population: Main Analysis Set with HAQ Score
Measure: Number; unit: participants
Groups:
- Improved: Clinically relevant improvement of HAQ-Score ≥0.3
- No Change: Other or no clinical relevant change of HAQ-Score
- Worse: Clinically relevant worsening of HAQ Score ≥0.3
Arm/Group | Improved | No Change | Worse
Number analyzed (Participants) | 253 | 366 | 76
participants
  Subgroup 1: Anti-CCP-/RF- (n=44) | 10 | 28 | 6
  Subgroup 2: Anti-CCP-/RF+ (n=19) | 2 | 17 | 0
  Subgroup 3: Anti-CCP+/RF- (n=45) | 14 | 29 | 2
  Subgroup 4: Anti-CCP+/RF+ (n=375) | 146 | 185 | 44
  Subgroup 5: Anti-CCP n.sp./RF+ (n=109) | 46 | 57 | 6
  Subgroup 6: Anti-CCP n.sp./RF- (n=29) | 9 | 13 | 7
  Subgroup 7: Anti-CCP+/RF n.sp. (n=19) | 8 | 7 | 4
  Subgroup 8: Anti-CCP-/RF n.sp. (n=2) | 0 | 1 | 1
  Subgroup 9: Seropositive n.sp. (n=17) | 6 | 9 | 2
  Subgroup 10: Anti-CCP and RF n.sp. (n=36) | 12 | 20 | 4
  Subgroup 1+6+8: seronegative (n=75) | 19 | 42 | 14
  Subgroup 2+3+4+5+7+9: seropositive (n=584) | 222 | 304 | 58

5. Secondary Outcome: Number of Participants Who Received Two Cycles With Clinically Relevant Changes in HAQ-Score at Last Visit During Therapy Compared to Baseline (Categorized)
Description: In the Subpopulation With Two Cycles, the HAQ score was categorized for 12 subgroups as Clinically relevant improvement of HAQ-Score ≥0.3, Other or no clinical relevant change of HAQ Score, or Clinically relevant worsening of HAQ Score ≥0.3. Subgroups are defined as Anti-Cyclic citrullinated peptide (CCP) and Rheumatoid factor (RF) negative (-), positive (+), or Non-specified (n.sp.) and Seropositive Non-specified (n.sp.), Seronegative, or Seropositive.
Time Frame: 24 weeks after starting Cycle 2
Population: Subpopulation With Two Cycles with HAQ Score
Measure: Number; unit: participants
Arm/Group | Improved | No Change | Worse
Number analyzed (Participants) | 233 | 243 | 83
participants
  Subgroup 1: Anti-CCP-/RF- (n=33) | 7 | 17 | 9
  Subgroup 2: Anti-CCP-/RF+ (n=11) | 4 | 6 | 1
  Subgroup 3: Anti-CCP+/RF- (n=36) | 8 | 18 | 10
  Subgroup 4: Anti-CCP+/RF+ (n=314) | 147 | 130 | 37
  Subgroup 5: Anti-CCP n.sp./RF+ (n=100) | 42 | 44 | 14
  Subgroup 6: Anti-CCP n.sp./RF- (n=17) | 3 | 6 | 8
  Subgroup 7: Anti-CCP+/RF n.sp. (n=14) | 10 | 3 | 1
  Subgroup 8: Anti-CCP-/RF n.sp. (n=2) | 1 | 1 | 0
  Subgroup 9: Seropositive n.sp. (n=10) | 5 | 4 | 1
  Subgroup 10: Anti-CCP and RF n.sp. (n=22) | 6 | 14 | 2
  Subgroup 1+6+8: seronegative (n=52) | 11 | 24 | 17
  Subgroup 2+3+4+5+7+9: seropositive (n=485) | 216 | 205 | 64

ADVERSE EVENTS:
Time Frame: 3 years, 6 months
Description: AEs which cannot be assigned to a Cycle due to missing/incomplete start date are counted in the Total column only
Groups:
- Total: During the entire trial
Arm/Group | Cycle 1 | Cycle 2 | Total
Serious Adverse Events (participants affected / at risk) | 144/1653 | 47/820 | 180/1653
Other Adverse Events (participants affected / at risk) | 0/1653 | 0/820 | 0/1653
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cycle 1 (N=1653) | Cycle 2 (N=820) | Total (N=1653)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 2
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 4 | 0 | 4
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 3
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 4 | 2 | 6
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 3 | 0 | 3
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1 | 3
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 2 | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0 | 1
Macular degeneration (Eye disorders) | 1 | 0 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0 | 2
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 1
Chest discomfort (General disorders) | 2 | 0 | 2
Chest pain (General disorders) | 2 | 1 | 3
Chills (General disorders) | 3 | 0 | 3
Death (General disorders) | 3 | 1 | 4
Device dislocation (General disorders) | 1 | 0 | 1
Drug effect decreased (General disorders) | 1 | 0 | 2
Drug ineffective (General disorders) | 1 | 0 | 1
Drug interaction (General disorders) | 1 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 1
Generalised oedema (General disorders) | 0 | 1 | 1
Hyperplasia (General disorders) | 1 | 0 | 1
Impaired healing (General disorders) | 1 | 1 | 2
Influenza like illness (General disorders) | 1 | 0 | 1
Infusion related reaction (General disorders) | 1 | 1 | 2
Local swelling (General disorders) | 1 | 0 | 1
Malaise (General disorders) | 1 | 0 | 1
Medical device complication (General disorders) | 0 | 1 | 1
Multi-organ failure (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1
Pain (General disorders) | 3 | 0 | 3
Pyrexia (General disorders) | 2 | 1 | 3
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Gallbladder cholesterolosis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 1
Antiphospholipid syndrome (Immune system disorders) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 4 | 0 | 4
Abscess (Infections and infestations) | 1 | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0 | 1
Acute endocarditis (Infections and infestations) | 1 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 1
Breast abscess (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 5 | 2 | 7
Cellulitis (Infections and infestations) | 2 | 1 | 3
Cranial nerve infection (Infections and infestations) | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 1
Encephalitis brain stem (Infections and infestations) | 1 | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 2
Herpes simplex (Infections and infestations) | 1 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 5 | 1 | 6
Infected cyst (Infections and infestations) | 1 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 1
Pneumococcal infection (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 11 | 2 | 13
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 2 | 0 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1 | 1
Viral infection (Infections and infestations) | 1 | 0 | 1
Accident (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 0 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 2 | 0 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Biopsy prostate (Investigations) | 1 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 1
Fibrin D dimer increased (Investigations) | 1 | 0 | 1
Prostatic acid phosphatase increased (Investigations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 | 1 | 6
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 7 | 4 | 10
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 2
Disturbance in attention (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 1
Sciatica (Nervous system disorders) | 2 | 0 | 2
Syncope (Nervous system disorders) | 1 | 3 | 4
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | 2
Depression (Psychiatric disorders) | 1 | 0 | 1
Nightmare (Psychiatric disorders) | 1 | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 0 | 1
Bladder tamponade (Renal and urinary disorders) | 1 | 0 | 1
Cystitis glandularis (Renal and urinary disorders) | 2 | 0 | 2
Renal artery stenosis (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Breast disorder (Reproductive system and breast disorders) | 1 | 0 | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Arterial repair (Surgical and medical procedures) | 1 | 0 | 1
Carpal tunnel decompression (Surgical and medical procedures) | 1 | 0 | 1
Cataract operation (Surgical and medical procedures) | 1 | 0 | 1
Elbow operation (Surgical and medical procedures) | 1 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 1 | 1 | 2
Hospitalisation (Surgical and medical procedures) | 2 | 0 | 2
Intervertebral disc operation (Surgical and medical procedures) | 1 | 0 | 1
Joint arthroplasty (Surgical and medical procedures) | 1 | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 1 | 2
Nasal septal operation (Surgical and medical procedures) | 0 | 1 | 1
Rotator cuff repair (Surgical and medical procedures) | 1 | 0 | 1
Shoulder operation (Surgical and medical procedures) | 1 | 0 | 1
Sinus operation (Surgical and medical procedures) | 0 | 2 | 2
Spinal fusion surgery (Surgical and medical procedures) | 1 | 1 | 2
Spinal operation (Surgical and medical procedures) | 0 | 1 | 1
Tendon operation (Surgical and medical procedures) | 0 | 1 | 1
Tendon sheath incision (Surgical and medical procedures) | 0 | 1 | 1
Circulatory collapse (Vascular disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Embolism arterial (Vascular disorders) | 0 | 1 | 1
Haematoma (Vascular disorders) | 1 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 2 | 0 | 2
Hypotension (Vascular disorders) | 3 | 0 | 3
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.